CLINICAL TRIAL: NCT00221715
Title: Randomised Study Comparing Prosthesis and Autologous Vein for Revascularisation With Above Knee Femoropopliteal Bypass.
Brief Title: Comparison of Two Lower Limb Bypass Types : Prosthesis Versus Autologous Vein
Acronym: REVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9248-01; 2000-006
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Arteritis; Diabetes
Keywords: arteritis; lower limb ischemia; femoropopliteal artery bypass; blood vessel prothesis implantation; saphenous vein; vascular permeability; doppler ultrasonography; randomized clinical trials; efficacy study
MeSH Terms: conditions — Arteritis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): bypass by autologous saphenous vein
  Interventions: Device: femoropopliteal artery bypass
- 2 (Active Comparator): bypass by dacron or PTFE Prosthesis
  Interventions: Device: femoropopliteal artery bypass

INTERVENTIONS:
Device: femoropopliteal artery bypass — Bypass by autologous saphenous vein
  Arms: 1
Device: femoropopliteal artery bypass — bypass by dacron or PTFE Prosthesis
  Arms: 2

SUMMARY:
When medical treatments fail, critical ischemia of the lower limb often leads to surgery, i.e. above knee femoro popliteal bypass. This bypass can be performed either with DACRON or PTFE prosthesis or with the autologous saphenous vein. Both technics are used but they have not been compared regarding bypass permeability and limb salvage. Thus, this study will compare the permeability rate of above knee femoro popliteal surgery whether performed with autologous vein versus prosthesis

DETAILED DESCRIPTION:
When medical treatments fail, critical ischemia of the lower limb often leads to surgery, i.e. above knee femoro popliteal bypass. This bypass can be performed with either DACRON or PTFE prosthesis or with the autologous saphenous vein. The principle disadvantages of prosthesis are their prejudged worse permeability and the risk of infection. Too few reliable randomised, multicentric studies in this indication comparing vein bypasses versus prosthesis bypasses have been conducted to firmly confirm the first argument. Thus, the purpose of this multicentric, randomised, national study is to compare, 5 years after surgery, the permeability rate of above knee femoropopliteal bypass with vein versus prosthesis. Primary and secondary permeability, permeability predictive factors, and leg salvage rate will also be assessed. One hundred enrolled patients with II to IV level leg arteritis will randomly be assigned to one of the surgery groups : vein or prosthesis (50 each). The recruiting period will last 3 years and a half, and the follow up 5 years for each patient. The main primary outcome, bypass permeability, will be assessed through Doppler ultrasonography during five years. Secondary endpoints, mortality and morbidity, will be evaluated during the clinical follow up. Permeability predictive factors, primary and secondary permeability, leg salvage will also be recorded. If the permeability rates are equivalent between prosthesis and vein, the use of prosthesis will be preferred as this surgery is easier and faster, and as it is important that the vein remains available for distal revascularisation (where it is more efficient) and for revascularisation of coronary arteries

ELIGIBILITY:
Inclusion Criteria:

* lower limbs arteritis : II to IV arteritis level, above knee femoro popliteal bypass indication
* signed informed consent

Exclusion Criteria:

* no contra indication to the use of prosthesis
* Available saphenous vein
* no major trophic trouble

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Bypass permeability 5 years after surgery, assessed trough Doppler ultrasonography | 5 years

SECONDARY OUTCOMES:
Mortality | 5 years
Morbidity | 5 years
permeability predictive factors (smoking habits, diabetes, hyperlipidemia, bypass diameter) | 5 years
Primary and secondary permeability | 5 years
leg salvage | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Midy, Professor, Principal Investigator — University Hospital, Bordeaux; Geneviève Chêne, Professor, Study Chair — University Hospital, Bordeaux